CLINICAL TRIAL: NCT05166356
Title: Describing the Determinants and Effects of Variation in the Adoption and Use of the NOHARM Pain Management Intervention Among Diverse Surgical Practices
Brief Title: Determinants and Effects in the Use of NOHARM Pain Management
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Andrea Cheville, Principal Investigator, Mayo Clinic
Other Study IDs: 21-007898; UH3AG067593-03 (NIH)
Record Dates: First submitted 2021-10-28; First posted 2021-12-21 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: A sample of patients who received the NOHARM intervention after their surgery.
- Care Team Members: Staff members who had patients on the NOHARM intervention

SUMMARY:
The objective of this study is to enrich the ongoing Non-pharmacological Pain Management After Surgery (NOHARM) pragmatic trial (NCT04570371) with a mixed methods analysis of patient and care team factors that affect the routine adoption, implementation, and meaningful and sustainable use of the NOHARM intervention.

DETAILED DESCRIPTION:
Aim 1: Explore differences in patient engagement with the NOHARM intervention, use of non-pharm modalities, and clinical outcomes by key patient demographics, including surgical procedure type, gender, and opioid abuse risk. This aim will provide information about patient characteristics that may better predict who will use and/or benefit from the NOHARM intervention and who will not.

Aim 2: Qualitatively explore determinants of patient-level factors contributing to their ability to effectively engage with the NOHARM intervention in a diverse subgroups that adopt and use the intervention as intended and those that do not, respectively. This aim will provide information that helps us explain why some patients tend to use and/or benefit from NOHARM and others do not.

Aim 3: Characterize, using mixed methods, the relative fidelity and sustainability of implementation of NOHARM among ambulatory and inpatient surgical practices and test for associations with patient engagement and clinical outcomes. This aim will provide information about the characteristics of care teams that tend to adopt and maintain use of the NOHARM intervention and those that do not. It will also provide information about whether care teams play an important role in prompting patients to engage with and benefit from the NOHARM intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for this study will be patients on the NOHARM trial registry (e.g., patients that were automatically assigned to receive the NOHARM intervention as part of their surgical care) and/or their charts and members of their care teams, including nurses, doctors, physical therapists, nurse practitioners and physician assistants, and medical assistants.

Exclusion Criteria:

* Individuals not on the NOHARM trial registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will all be patients who received the NOHARM intervention for a recent surgery.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Aim 1 | 3 months post-surgery
  Characteristics of high and low fidelity users of the intervention
Determinants of patient engagement with the intervention | 3 months post-surgery
  Measured by the NOHARM patient interview guide that asks the participant to list determinants for non-medication options of managing pain
Sustainability of the NOHARM intervention | 3 months post-surgery
  Assessed using the Clinical Sustainability Assessment Tool (CSAT) that is a structured assessment of current capacity for sustainability across a range of specific organizational and contextual factors. Responses from the care team for this survey identify sustainability strengths and challenges. Questions use a scale of 1=to little or not extent and 7 = to a very great extent; scores are averaged for a total score with lower average scores indicating areas where practice capacity for sustainability could be improved.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cheville, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minteer SA, Audeh CM, Tofthagen C, Sheffield KE, Cutshall SM, Tilburt JC, Cheville AL. Patients' peri-operative experiences with non-pharmacologic pain care techniques: a secondary qualitative analysis of the NOHARM trial. BMC Complement Med Ther. 2025 Oct 17;25(1):388. doi: 10.1186/s12906-025-05141-0. PMID 41107758
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT05166356/Prot_007.pdf